CLINICAL TRIAL: NCT03406637
Title: Combined Prospective / Retrospective, Open, Non-randomized, Non-interventional Post Market Clinical Follow-Up of the BPK-S Integration System (Co28Cr6Mo) Used for Primary Total Knee Replacement
Brief Title: Combined Prospective and Retrospective Post-Market Follow Up of the 'BPK-S Integration' UC as Primary Implant in the Variant CoCr
Status: Completed | Type: Observational
Sponsor: Peter Brehm GmbH (Industry)
Collaborators: P.R.I.S.M.A.-CRO (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2016-01-BPK-S
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis, Knee; Joint Instability
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Instability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BPK-S Integration — primary total knee endoprosthesis

SUMMARY:
Patients who received a total knee endoprosthesis BPK-S Integration between 2011 and 2013 will be invited to participate in this PMCF study provided sufficient source data documentation is available regarding preoperative, intraoperative and early postoperative follow-up assessments.

Only patients providing written informed consent prior to any study data collection can take part in the study.

Preoperative, intraoperative and early postoperative data (3 months, 1 year and 2 years after implantation) will be collected retrospectively. Additional long-term follow-up of one visit (year 7 after implantation) will be documented prospectively.

Only parameters assessed in clinical standard care for follow-up (implant control) visits will be collected for this PMCF study.

Radiological assessment of the implanted prosthesis will only be conducted if medically indicated according to the investigator. No additional study related assessment will be performed.

Only anonymized data will be used in this observational study to protect patient privacy. No personally identifiable information will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients that received a total primary knee endoprosthesis BPK-S Integration (Co28Cr6Mo) between 2011 and 2013
* Patients that agree to participate and give written informed consent to the anonymized retrospective and prospective data collection within the study

Exclusion Criteria:

No study specific exclusion criteria are defined for this PMCF study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that received a BPK-S Integration in the variant CoCr as primary total knee endoprosthesis between 2011 and 2013 implanted by the investigator
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Patient relevant benefit after 5 years | 7 years
  improvement of KSS-Score by at least one category as compared to preoperative basic assessment

SECONDARY OUTCOMES:
Safety parameters | 7 years
  Incidents that require reporting to the competent authority and complications during and after surgery as documented in source documentation
Patient relevant benefit as measured by American Knee Society Score | 1 year
  improvement of KSS-Score as compared to preoperative basic assessment
Implant Loosening Number | 7 years
  Number of implant loosening due to quality issues with the implant
Implant Loosening Reason | 7 years
  Reason for implant loosening due to quality issues with the implant
Revision Number | 7 years
  Number of revisions, if required
Revision Reason | 7 years
  Reason for revision, if required
Surgery Parameters | Day 0 = day of surgery
  Evaluation of surgery time as documented in the surgical report
Surgery Parameters | Day 0 = day of surgery
  Evaluation of tourniquet time as documented in the surgical report

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Centre Hospitalier de Wallonie picarde - CHwapi A.S.B.L, Tournai
  - Medical Center Tournai, Tournai